CLINICAL TRIAL: NCT00459771
Title: Prospective, Randomized, Pharmacological Intervention Study; Evaluating Effect of the Angiotensin II-receptor (AT1) Blocker Candesartan vs Placebo in Prevention of Trastuzumab-associated Cardiotoxicity in Patients Treated With Trastuzumab
Brief Title: Evaluating the Effect of Candesartan vs Placebo in Prevention of Trastuzumab-associated Cardiotoxicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06HER; 2006-001707-11 (EudraCT Number)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: angiotensin II-receptor (AT1) blocker; prevention; trastuzumab; cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Candesartan (Active Comparator): Candasartan
  Interventions: Drug: AT1 blocker candesartan

INTERVENTIONS:
Drug: AT1 blocker candesartan — AT1 blocker candesartan, 32 mg oral QD
  Arms: Candesartan
Drug: Placebo — Placebo, 32 mg, oral QD
  Arms: Placebo

SUMMARY:
Evaluating the effect of the angiotensin II-receptor (AT1) blocker candesartan vs placebo in prevention of trastuzumab-associated cardiotoxicity in patients with primary breast cancer treated with trastuzumab.

DETAILED DESCRIPTION:
Prospective, randomized pharmacological intervention study

Primary objectives:

- to determine whether concurrent ATII-antagonist treatment can prevent trastuzumab-related cardiotoxicity, defined as a decline in LVEF of more than 15% or a decrease to an absolute value <45%

Secondary objectives:

* To determine if 'Brain Natriuretic Peptide' (NT-proBNP) and troponin T can be used as surrogate marker in the monitoring of trastuzumab-associated cardiotoxicity
* To determine genetic variability in relevant genes such as the HER2 gene (by assessing single nucleotide polymorphisms [SNPs] in the kinase domain) and explore any correlations with trastuzumab induced cardiotoxicity 3) To determine the reversibility of a decrease in left ventricular ejection fraction (LVEF) associated with trastuzumab treatment

Arm I : placebo Arm II : AT1 blocker candesartan (32 mg/day; run in 16 mg during week 1)

Randomization: before chemotherapy treatment period. Study period: chemotherapy period, trastuzumab treatment period 26 weeks follow up after discontinuation of trastuzumab treatment and thereafter 1 month follow-up after end of placebo or AT1 blocker.

Candesartan treatment will start the same day as the first infusion of trastuzumab and will continue up to 26 weeks after the end of treatment with trastuzumab.

Women with primary HER2 positive breast cancer who are considered for adjuvant systemic treatment with anthracycline containing chemotherapy and trastuzumab.

Before start of anthracycline treatment:

* Medical history, physical examination
* New York Heart Association (NYHA) score
* Cardiac questionnaire
* Electrocardiogram
* MUGA scan
* Laboratory assessments; hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, sodium, potassium, calcium, thyroid stimulating hormone, glucose, cholesterol, bilirubin, alkaline phosphatase, ASAT/ALAT, LDH, albumin, NT-proBNP, troponin T analysis
* Pregnancy test
* Genotype analysis

Every chemotherapy cycle

- Laboratory assessments; hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, sodium, potassium, calcium, glucose, bilirubin, alkaline phosphatase, ASAT/ALAT, LDH, albumin, (NT-proBNP, troponin T analysis)

Before start of trastuzumab treatment:

* Physical examination
* New York Heart Association (NYHA) score
* Cardiac questionnaire
* Electrocardiogram
* MUGA scan
* Laboratory assessments; hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, sodium, potassium, calcium, glucose, bilirubin, alkaline phosphatase, ASAT/ALAT, LDH, albumin, NT-proBNP, troponin T analysis

After 3, 6 and 9 months trastuzumab:

* Physical examination
* New York Heart Association (NYHA) score
* Cardiac questionnaire
* MUGA scan
* Laboratory assessments; hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, sodium, potassium, calcium, glucose, bilirubin, alkaline phosphatase, ASAT/ALAT, LDH, albumin, NT-proBNP, troponin T analysis

After 1 year trastuzumab, 26 weeks after the last trastuzumab administration:

* Physical examination
* New York Heart Association (NYHA) score
* Cardiac questionnaire
* Electrocardiogram
* MUGA scan
* Laboratory assessments; hemoglobin, hematocrit, white blood cell count, platelet count, serum creatinine, sodium, potassium, calcium, glucose, bilirubin, alkaline phosphatase, ASAT/ALAT, LDH, albumin, NT-proBNP, troponin T analysis

The primary endpoint of the study is the deterioration of the cardiac function defined as a decline in LVEF of 15% or more to an absolute value below 45% during the year with trastuzumab.

From previous studies it is estimated that about 30% of the patients treated with trastuzumab will show deterioration of LVEF.

A total of 200 patients will receive trastuzumab and candesartan or trastuzumab and placebo in this double blind placebo-controlled study. The number of patients randomized (= before chemotherapy period) for this trial shall be more than 200 as a small number of patients might drop out before start of therapy with trastuzumab. This number cannot exactly be determined beforehand.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years
* WHO: ≤ 2
* Strongly HER2-positive breast cancer, defined as an immunohistochemistry score of 3+ using the HercepTestTM, or gene amplification by fluorescence in situ hybridization, or chromogenic in situ hybridization (CISH).
* Serum creatinine <140 umol/l or creatinine clearance > 50 ml/min (by Cockcroft-Gault formula)
* Thyroid stimulating hormone between 0.5-3.9 MU/l
* Blood pressure systolic ≥ 140 mmHg and diastolic ≥ 90 mmHg is acceptable at randomization. However prior to the first administration of trastuzumab blood pressure should be regulated and should be systolic ≥ 100 mmHg and ≤ 180 mmHg and diastolic ≥ 60 mmHg and ≤ 100 mmHg. (blood pressure should be regulated according to the guidelines of appendix 5)
* LVEF ³ 50% assessed by multigated angiography (MUGA) or cardiac ultrasound
* Adjuvant regimen: trastuzumab start ≥ 3 weeks after day 1 of the last anthracycline chemotherapy cycle
* Trastuzumab treatment according to standard medical care
* Written informed consent to participate in the study

Exclusion Criteria:

* Prior anthracycline chemotherapy regimen or anti-HER2 therapy, or other prior biologic or immunotherapy for breast cancer treatment or any malignancy
* Previous malignancy requiring chemotherapy or radiotherapy
* Uncontrolled serious concurrent illness
* Patients with New York Heart Association (NYHA) class II/III/IV congestive heart failure
* Myocardial infarction < 6 months before randomization
* Treatment with ACE inhibitor, ATII blocker, or lithium. Patients treated with ACE inhibitor, or ATII blocker can switch (after randomization and during the chemotherapy period) to alternative antihypertensive therapy; see appendix 5.
* History of hypersensitivity to the study medication
* Pregnancy or breast feeding

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The occurrence of cardiotoxicity, defined as a decline in LVEF (MUGA) of more than 15% or a decrease of less than 15% to an absolute value below 45%. | during 1 year trastuzumab therapy and during 26 weeks after discontinuation of trastuzumab

CONTACTS AND LOCATIONS:
Overall Officials: J.H.M. Schellens, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (19):
- Netherlands (19):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - The Netherlands Cancer Institute, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Deventer Ziekenhuis, Deventer
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Groningen
  - University Medical Center Groningen, Groningen
  - Ziekenhuis de Tjongerschans, Heerenveen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Hospital, Nijmegen
  - UMC St. Radboud, Nijmegen
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo
  - Streekziekenhuis Koningin Beatrix, Winterswijk
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Boekhout AH, Gietema JA, Milojkovic Kerklaan B, van Werkhoven ED, Altena R, Honkoop A, Los M, Smit WM, Nieboer P, Smorenburg CH, Mandigers CM, van der Wouw AJ, Kessels L, van der Velden AW, Ottevanger PB, Smilde T, de Boer J, van Veldhuisen DJ, Kema IP, de Vries EG, Schellens JH. Angiotensin II-Receptor Inhibition With Candesartan to Prevent Trastuzumab-Related Cardiotoxic Effects in Patients With Early Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2016 Aug 1;2(8):1030-7. doi: 10.1001/jamaoncol.2016.1726. PMID 27348762